CLINICAL TRIAL: NCT06907472
Title: Integrating Diabetes Care Into Primary Healthcare Centers in Abuja, Nigeria: A Pilot Study
Brief Title: Diabetes Management for Primary Healthcare Centers.
Acronym: DM4PHC-pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Abuja (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Northwestern University (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ikechukwu Anthony Orji, Post-Doctoral Research Fellow, University of Abuja
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UATH/HREC/PR/505; D43TW011976 (NIH); FHREC/2024/01/190/06-08-24 (Other: FCT Health Research Ethics Committee)
Record Dates: First submitted 2025-03-14; First posted 2025-04-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Integrating Diabetes care; Primary Healthcare Center; pilot study; Abuja; Nigeria
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study is a single-arm pilot trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm diabetes management in Primary Healthcare Centers [PHCs] (Experimental): Single-arm diabetes treatment in two PHCs. The two PHCs will implement a contextually and culturally adapted package based on the WHO HEARTS-D package for screening, diabetes diagnosis, patient education, and treatment using a HEARTS-D-adapted treatment protocol.
  Interventions: Drug: Protocol-based treatment

INTERVENTIONS:
Drug: Protocol-based treatment — PROTOCOL:
  Step 1: Metformin 500 mg daily Step 2: Metformin 1000 mg daily Step 3: Metformin 1000 mg twice daily Step 4: Metformin 1000 mg twice daily + glibenclamide 5 mg daily Step 5: Metformin 1000 mg twice daily + glibenclamide 5 mg twice daily
  Other Names: 1. Metformin 500mg [brand; Diamet 500mg by MAY & BAKER Nigeria PLC] 2. Glibenclamide 5mg [brand; Diatab 5mg by MAY & BAKER Nigeria PLC]

SUMMARY:
The purpose of this study, "Integrating diabetes care into Primary Healthcare Centers (PHCs) in Abuja, Nigeria: a pilot study," is to screen, diagnose, treat, and educate diabetes patients in two selected PHCs in Abuja. This single-arm pilot trial will test the feasibility of integrated diabetes care, measure the implementation outcomes, and explore the effectiveness of the strategy bundle using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

DETAILED DESCRIPTION:
The pilot study involves the use of non-physician health workers (e.g., community health extension workers [CHEWs], nurses, and laboratory technicians) to implement a diabetes care program in alignment with the HEARTS diabetes-specific module, also known as HEARTS-D. The study adapted strategies from the Transforming Hypertension Treatment in Nigeria (HTN) Program, originally based on the Kaiser Permanente Northern California hypertension program and HEARTS technical package. The adapted intervention is informed by experience from the successful HTN program and findings from the investigators' formative assessment for this diabetes integration in the PHC setting.

The investigators used an adapted Service Availability and Readiness Assessment (SARA) instrument for the formative assessment and evaluated the PHC's availability and readiness for diabetes care across various domains. These domains include staffing, training, equipment, medications, clinical guidelines, health management information systems, and diabetes care services. The formative study also assessed health workers' knowledge, attitudes, and practices related to diabetes care and explored barriers and facilitators of implementing diabetes treatment programs at the PHC setting. The findings from the formative work informed the development and adaptation of strategies for this pilot implementation. The investigators are leveraging the available non-physician health workers and paper-based health management information systems, strengthening diabetes screening and counselling services, providing adequate training and re-training of health workers to provide comprehensive diabetes care services, providing diabetes education materials and job aids, and improving access to diabetes medications. The strategy is designed to overcome modifiable barriers at patient and system levels in the cascade of care for diabetes care at the PHC setting in Nigeria.

This pilot study will deliver a multi-level implementation package for diabetes care, which includes:

1. Healthy lifestyle counseling on clinic visits (Patient level).
2. Simplified treatment protocol for diabetes management (National policy level).
3. Access to functioning glucometers, test strips, and essential medicines (Health systems level).
4. Team-based care and trained Community health extension workers/nurses to provide Diabetes management and follow up care (Health workers & National Policy level).
5. Information system to support performance and quality reporting and Health facility improvement (Health facility level).
6. Diabetes patient registry and empanelment (Health system level).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Uncomplicated type 2 diabetes mellitus

Exclusion Criteria:

* Minors (younger than 18 years),
* Type 1 diabetes mellitus
* Prisoners
* Other detained individuals
* Severe hypertension (SBP ≥180 mmHg and DBP ≥ 110 mmHg)
* Prior history of complications: stroke, heart failure, chronic kidney disease, diabetic foot ulcer.
* Pregnant women.
* Older patients above 60 years of age with uncontrolled plasma glucose at the maximum dose of metformin (2 g/day) and maximum dose of glibenclamide (5mg/day) at entry to the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Reach (Recruitment rate): defined as the proportion of patients enrolled per month per the monthly recruitment target. | Six months.
  BENCHMARK: Achieving 50% of the monthly recruitment target of 18 participants per month.
  MEASUREMENT: Number of eligible patients recruited by participating PHCs per month divided by Monthly recruitment target x 100%
Adoption (adherence to protocol): defined as the proportion of diagnosed patients with diabetes started on treatment. | Six months.
  BENCHMARK: Achieving 80% treatment rate MEASUREMENT: The number of diagnosed patients with diabetes started on treatment divided by the total number of enrolled diabetes patients in the study x 100%.
Maintenance (retention rate): defined as the proportion of patients who complete the six-month final visit of the implementation phase | Six months.
  BENCHMARK: Achieving a 50% retention rate. MEASUREMENT: The total number of patients who complete the six-month final visit divided by the total number of enrolled patients during the six months of implementation x 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Ikechukwu A. Orji, MBBS, PhD, Principal Investigator — University of Abuja; Dike B. Ojji, MBBS, PhD, Study Chair — University of Abuja; Lisa R. Hirschhorn, MD, MPH, Study Director — Northwestern University Chicago
Locations (2):
- Nigeria (2):
  - Kagini PHC, Abuja Municipal Area council (AMAC), Abuja, Federal Capital Territory
  - Deidei PHC, Bwari Area Council, Abuja, Federal Capital Territory

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared through NHLBI BioLINCC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 1 year of study's conclusion.
Access Criteria: Access to study data will be managed through NHLBI BioLINCC.
URL: https://redcap.uniabuja.edu.ng/redcap_v13.0.1/index.php?pid=203&__record_cache_complete=1

REFERENCES:
- [Result] Baldridge AS, Aluka-Omitiran K, Orji IA, Shedul GL, Ojo TM, Eze H, Shedul G, Ugwuneji EN, Egenti NB, Okoli RCB, Ale BM, Nwankwo A, Osagie S, Ye J, Chopra A, Sanuade OA, Tripathi P, Kandula NR, Hirschhorn LR, Huffman MD, Ojji DB. Hypertension Treatment in Nigeria (HTN) Program: rationale and design for a type 2 hybrid, effectiveness, and implementation interrupted time series trial. Implement Sci Commun. 2022 Aug 2;3(1):84. doi: 10.1186/s43058-022-00328-9. PMID 35918703
- [Result] Orji IA, Baldridge AS, Omitiran K, Guo M, Ajisegiri WS, Ojo TM, Shedul G, Kandula NR, Hirschhorn LR, Huffman MD, Ojji DB. Capacity and site readiness for hypertension control program implementation in the Federal Capital Territory of Nigeria: a cross-sectional study. BMC Health Serv Res. 2021 Apr 9;21(1):322. doi: 10.1186/s12913-021-06320-8. PMID 33836719
- [Result] Orji IA, Baldridge AS, Ikechukwu-Orji MU, Banigbe B, Eze NC, Chopra A, Omitiran K, Iyer G, Odoh D, Alex-Okoh M, Reng R, Hirschhorn LR, Huffman MD, Ojji DB. Evaluation of Primary Healthcare Centers' Service Availability and Readiness for Implementing Diabetes Care in Abuja, Nigeria: A Cross-Sectional, Formative Assessment. Res Sq [Preprint]. 2024 Mar 26:rs.3.rs-3959541. doi: 10.21203/rs.3.rs-3959541/v1. PMID 38585872
- See also: University of Abuja REDCap link to participant data set. — https://redcap.uniabuja.edu.ng/redcap_v13.0.1/index.php?pid=203&__record_cache_complete=1
- Available data/document: Individual Participant Data Set — https://redcap.uniabuja.edu.ng/redcap_v13.0.1/index.php?pid=203&__record_cache_complete=1 — University of Abuja REDCap link to participant data set.